CLINICAL TRIAL: NCT03479775
Title: The Role of Muscle Function as a Potential Risk and/or Protective Factor for Traumatic Knee Injury in Youth Female Athletes
Brief Title: Muscle Function and Traumatic Knee Injury in Sports
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 929-13
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: ACL Injury; Meniscus Lesion; Cartilage Injury; Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Youth female athletes with poor muscle function: Youth female athletes (floorball, football and handball) with assessed poor muscle function at baseline.
- Youth female athletes with good muscle function: Youth female athletes (floorball, football and handball) with assessed good muscle function at baseline.

SUMMARY:
The aims of the project are to 1) evaluate different aspects of muscle function and its role as a potential risk and/or protective factor for traumatic knee injury in youth female athletes; 2) develop and evaluate a battery of muscle function tests, easily used and requiring minimal equipment, to be applied as an on-the-field screening tool to detect muscle function deficiencies and monitoring youth female athletes at high risk of traumatic knee injury.

A prospective cohort design will be used, including approximately 100 female athletes (age 15-19) from Swedish senior sports high schools who are involved in high risk sports (soccer, handball, floorball and basket). A test battery for muscle function has been developed consisting of 11 tests that previously have been used for the assessment of muscle function. The tests will be instructed and supervised by educated test leaders. Measurements will take place at the athletes' school and carried out during the first semester (autumn 2017 and 2018). Data on injury surveillance and exposure (hours of match and training participation) will be collected prospectively over two years using a web-designed registration form. All athletes will on a weekly basis report their hours of training, minutes of match play and all time-loss injuries occurring during sport activity. Details on injury mechanism and diagnosis will be collected by each school's medical staff. The present study will contribute new knowledge on the role of muscle function and develop and evaluate a battery of muscle function tests to be used as an on-the-field screening tool for monitoring youth female athletes at high risk of traumatic knee injury.

DETAILED DESCRIPTION:
A prospective cohort design will be used for the present study comprising approximately 100 (determined by power analysis) female athletes (age 15-19) from Swedish senior high schools who are involved in high risk sports (soccer, handball, floorball and basket). The study started autumn 2017 with assessment of muscle function at baseline, instructed and supervised by two test leaders. Before the test session the athlete will be informed and tutored about the injury and exposure registration procedure. Measurements takes place in a secluded room at the athletes' school and will be carried out during the first semester (autumn 2017, 2018, 2019 and 2020). Data relating to sport affiliation, number of years of specific sport training, the number of training hours per week and her/his training routines, level of competition and participation in other sports, age, body weight and height will also be conducted using a questionnaire. After the baseline assessment, the athletes will participate in a continuous web based prospective injury registration protocol and be followed for two years.

Outcome measures Data on injury surveillance and exposure (hours of match and training participation) will be collected prospectively over two years using a web-designed (REDCap Software) registration form. All athletes will on a weekly basis report their hours of training, minutes of match play and all time-loss injuries occurring during sport activity. Details on injury mechanism, nature, and diagnosis will be collected by each school's medical staff. The outcome of interest is a traumatic knee injury, i.e., ACL or other ligament injury, meniscal, cartilage damage or fracture, diagnosed by physical examination and/or MRI, arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Female high-school athlete
* age 15-19 y
* must play soccer, handball, floorball or basketplayer

Exclusion Criteria:

* illness, which might affect the test results
* injury to the lower extremity at the time of baseline data collection -

Ages: 15 Years to 19 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Female athletes (age 15-19) from Swedish senior high schools who are involved in high risk sports (soccer, handball, floorball and basket).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of traumatic knee injury | 2 years
  Traumatic knee injury will be assessed by a web-designed (REDCap Software) registration form
Muscle strength testing | Collected during 2 month at 1 session
  Muscle strength will be assessed using an isometric handheld dynamometer (Commander Echo, JTECH Medical, Salt Lake City, Utah, USA)
Muscular endurance and neuromuscular tests | Collected during 2 month at 1 session
  Muscular endurance and neuromuscular tests will be video-recorded using the Coach Eye app for smart phone

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Ryman Augustsson, Study Director — Lunds University
Locations (1):
- Sofia Ryman Augustsson, Kalmar, WV, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT03479775/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT03479775/SAP_001.pdf